CLINICAL TRIAL: NCT06985056
Title: Reducing Symptom Burden Through Physical Exercise in Melanoma Patients Under Immuno- or Targeted Therapy
Brief Title: Reducing Symptom Burden Through Physical Exercise in Melanoma Patients
Acronym: RESPECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Miriam Götte, PD Dr., Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RESPECT
Record Dates: First submitted 2025-05-08; First posted 2025-05-22 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Malignant Melanoma
Keywords: Exercise; Fatigue; Physical Activity; Checkpoint Inhibitors; BRAF/MEK Inhibitors; Melanoma; Quality of Life
MeSH Terms: conditions — Melanoma; Motor Activity; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): The supervised progressive endurance and resistance exercise program will be conducted twice per week online in small groups and will be guided by a sports scientist over a period of 12 weeks. All sessions will start with a warm-up, transitioning to endurance training, followed by strength exercises and finishing with a cool-down, and will take approximately 60 minutes. The moderate-to-high-intensity endurance training will be performed at the beginning of each training session for 15 minutes in the range of the ventilatory threshold 1 (VT1), which was obtained during the baseline cardiorespiratory exercise test. The moderate-to-high-intensity progressive resistance training and bodyweight regime will include 6 exercises that target major upper and lower body muscle groups as well as trunk exercises. Resistance exercise includes free weight, resistance bands, and bodyweight workouts.
  Interventions: Behavioral: Supervised 12-week Resistance and Endurance Exercise Program
- Control Group (No Intervention): Control group will receive usual care without an exercise program. After the final endpoint assessment, patients randomized into the control group will be offered the opportunity to participate in an exercise program conducted by the Sports and Exercise Therapy Group at WTZ Essen.

INTERVENTIONS:
Behavioral: Supervised 12-week Resistance and Endurance Exercise Program — 60 Minute home-based and supervised endurance, resistance and coordination training 2x/week for 12 weeks, self-administered 20 minute home-based multimodal training 1x/week
  Arms: Exercise Intervention

SUMMARY:
The aim of the clinical trial is to determine whether regular exercise can reduce fatigue in adult patients with stage IIb-IV melanoma undergoing immunotherapy or targeted therapy. Additionally, we will investigate whether a supervised exercise program improves patients' quality of life, cognitive skills, and physical fitness compared to a control group without structured exercise. We will also examine other health outcomes and various blood parameters, such as interleukins and metabolites, to understand how regular activity can affect metabolism and immune function.

After the initial assessment at the clinic, patients will be randomly assigned to two groups. Those in the intervention group will participate in a 12-week exercise program, which includes a 60-minute personalized and supervised online training session twice a week. In weeks 3, 6, and 9, one training session will be held at the clinic. Furthermore, patients in the intervention group are encouraged to complete a self-administered 20-minute exercise session once a week. The control group will not receive a supervised exercise program. Following the 12-week intervention period, another assessment will be conducted at the clinic. All patients will then enter a 6-week follow-up phase, during which neither group will receive supervised exercise training. After this follow-up phase, a final assessment of all outcomes will take place at the clinic.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years with malignant melanoma (Stage IIb - IV) receiving adjuvant immuno- or targeted therapy
* patients already on the same treatment protocol for at least 3 months
* sufficient knowledge of German
* completed and signed written consent form and completed medical history form
* medical clearance for the exercise program and performance diagnostics
* ability to participate in the exercise program
* willingness to visit the study hospital for training sessions and examinations

Exclusion Criteria:

* confirmation of contraindications for physical exercise by the attending physician (e.g. fracture risk in the case of bone metastases)
* untreated, symptomatic, known brain metastases
* severe neurological or cardiac impairment according to ACSM criteria
* confirmation of respiratory insufficiency by the attending physician
* life expectancy less than 3 months
* physical or mental conditions that would not allow implementation of the exercise program or study protocol
* excessive physical activity (i.e. >150 minutes/week of moderate to intense physical activity and systematic intense strength/endurance training at least twice a week for one hour)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Fatigue | From baseline assessment to the end of treatment at 12 weeks
  Fatigue will be assessed with the validated 40-item Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F, version 4). It includes four multi-item functional scales (physical, social, emotional and functional well-being) and a multi-item symptom scale (fatigue).

SECONDARY OUTCOMES:
Fatigue | From the end of treatment to follow-up assessment at 18 weeks
  Fatigue will be assessed with the validated 40-item Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F, version 4). It includes four multi-item functional scales (physical, social, emotional and functional well-being) and a multi-item symptom scale (fatigue).
Quality of life of melanoma patients | From baseline assessment to the end of treatment at 12 weeks, from the end of treatment to follow-up assessment at 18 weeks
  Quality of Life (QoL) will be assessed with the validated 51-item Functional Assessment of Cancer Therapy - Melanoma (FACT-M, version 3). It includes four multi-item functional scales (physical, social, emotional and functional well-being) and a multi-item disease-specific subscale.
Physical Activity Behaviour | From baseline assessment to the end of treatment at 12 weeks, from the end of treatment to follow-up assessment at 18 weeks
  Physical Activity (PA) behaviour in the domains of activity at work, during leisure time, and exercise activity will be assessed via a standardized and validated questionnaire, the Physical activity and Sports activity Questionnaire (Bewegungs- und SportAktivitätsfragebogen (BSA, version 3.0)).
Strength of large muscle groups | From baseline assessment to the end of treatment at 12 weeks, from the end of treatment to follow-up assessment at 18 weeks
  Muscle strength will be assessed via 5-repetition-maximum strength test for large muscle groups. The protocol includes leg press, bench press, and lat pulldown
Cardiopulmonary fitness | From baseline assessment to the end of treatment at 12 weeks, from the end of treatment to follow-up assessment at 18 weeks
  Cardiopulmonary fitness will be measured by assessing maximal aerobic capacity (VO2peak) via a cycling test with a protocol starting at 20 watts and increasing by 10 watts every minute until the patient reaches volitional exhaustion. To control for test validity, gas exchange will be measured using a breath-by-breath gas analysis system which will be calibrated according to the manufacturer's instructions before each test. Patients' safety will be monitored. Blood pressure will be measured prior, during and after testing. The criteria for exhaustion will be fulfilled if two out of five of the following criteria are valid: (1) Borg scale > 16; (2) peak heart rate ± 10% of age-appropriate reference value; (3) oxygen saturation <88%; (4) patient is not able to maintain 60rpm and/or (5) respiratory exchange ratio (RER) > 1.1. Exercise will be terminated prematurely in the case of severe dyspnea or excessive blood pressure increase (≥250 mmHg systolic and/or ≥110 mmHg diastolic).
Cognitive Performance | From baseline assessment to the end of treatment at 12 weeks, from the end of treatment to follow-up assessment at 18 weeks
  The Montreal Cognitive Assessment (MoCA, version 8.1, 8.2 and 8.3) is a validated, highly sensitive tool for early detection of mild cognitive impairment. It generates a total score and six domain-specified index scores: (1) Memory, (2) Executive Functioning, (3) Attention, (4) Language, (5) Visuospatial, (6) Orientation. Three different versions are used across three different measurement timepoints to avoid practice-related improvements in test scores.
Body composition | From baseline assessment to the end of treatment at 12 weeks, from the end of treatment to follow-up assessment at 18 weeks
  Body composition will be assessed via bioelectrical impedance analysis (BIA). Body composition analysis includes (1) fat mass (FM); (2) fat-free mass (FFM); (3) body cell mass (BCM); (4) relative amount of external cell water (ECW%); (5) total body water (TBW); (6) intra cellular water (ICW); (7) appendicular skeletal muscle mass (ASMM) and (8) appendicular skeletal muscle mass index (ASMI). It also includes measurement of patients' weight and height, and the corresponding BMI.
Weight | From baseline assessment to the end of treatment at 12 weeks, from the end of treatment to follow-up assessment at 18 weeks
  Weight will be assessed in kilograms.
Height | From baseline assessment to the end of treatment at 12 weeks, from the end of treatment to follow-up assessment at 18 weeks
  Height will be assessed in meters.
BMI | From baseline assessment to the end of treatment at 12 weeks, from the end of treatment to follow-up assessment at 18 weeks
  Weight and height will be combined to report BMI in kg/m².
Blood pressure at rest | From baseline assessment to the end of treatment at 12 weeks, from the end of treatment to follow-up assessment at 18 weeks
  Assessment of blood pressure (diastolic and systolic) at rest will be conducted prior to exercise testing
Resting heart rate | From baseline assessment to the end of treatment at 12 weeks, from the end of treatment to follow-up assessment at 18 weeks
  Assessment of resting heart rate will be conducted prior to exercise testing.
Side effects/ symptoms | From baseline assessment to the end of treatment at 12 weeks, from the end of treatment to follow-up assessment at 18 weeks
  Evaluation of side effects or symptoms will be done via patient reported outcomes using Common Terminology Criteria for Adverse Events (PRO- CTCAE). Therefore, a standardized questionnaire containing 10 items covering most common therapy related symptoms such as (1) nausea; (2) vomiting; (3) diarrhea; (4) shortness of breath; (5) cough; (6) rash; (7) itching; (8) joint pain; (9) muscle pain; (10) decreased libido will be completed.
Response to therapy | From baseline assessment to the end of treatment at 12 weeks, from the end of treatment to follow-up assessment at 18 weeks
  Blood samples will be collected at all assessment time points in the clinic. Response will be assessed by determining the common melanoma tumor markers S100 and lactate dehydrogenase (LDH).
Blood parameters | From baseline assessment to the end of treatment at 12 weeks, from the end of treatment to follow-up assessment at 18 weeks
  Blood samples will be collected at all assessment time points in the clinic. Analysis of blood parameters will be conducted after the last patients' study completion to avoid batch effect in blood analysis. The following blood parameters will be analyzed: (1) metabolites (glucose, lactate, triglycerides, pyruvate, glycogen, alanine, PEP, citrate, succinate, fumarate, malate); (2) interleukins (IL-2, IL-6, IL-8, IL-10, IL-12, IL-15, IL-17, IL-23); (3) differential blood count (lymphocytes, haemoglobin levels)
Adherence | During the intervention phase
  Evaluation of patients' ability to fulfill the exercise prescription through assessment of absolute and relative numbers of completed versus planned exercise sessions.
Assessment of Safety | During the intervention phase
  Documentation of adverse events (AEs or SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Götte, PD Dr., Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: No